CLINICAL TRIAL: NCT03886766
Title: Bioavailability Mechanistic Study of Hot-Melt-Extruded Amorphous Solid Dispersions
Brief Title: Bioavailability Mechanistic Study of Hot-Melt Extruded Amorphous Solid Dispersions
Acronym: BEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-00282; ex18Huwyler
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2021-04

CONDITIONS: Biological Availability; Amorphous Solid Dispersions
Keywords: amorphous solid dispersion; Plasma concentration-time profile; Hot-Melt Extrusion

STUDY DESIGN:
Intervention Model Description: The intervention consists of a single oral administration of 3 different formulations containing Efavirenz as model drug tracer in sub-therapeutic doses:
  1. Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, oral administration (product 1)
  2. Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, homogenized to drug rich particles, oral administration (product 2)
  3. Efavirenz solution, 3 mg, oral administration (product 3) On the first visit, subjects will be randomized into three groups, starting with the ingestion of study product 1, 2, or 3 with subsequent collection of blood samples for 72 hours. After a wash out period of two weeks, participants will repeat the procedure in phase B with ingestion of the subsequent study product. After a second wash out the participants will receive the last study product in study phase C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence 1,2,3 (Experimental): Period A/ Visit 2: Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, oral administration (product 1) Period B/ Visit 6: Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, homogenized to drug rich particles, oral administration (product 2) Period C/ Visit 10: Efavirenz solution, 3 mg, oral administration (product 3)
  Interventions: Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz; Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz homogenized to drug rich particles; Drug: Efavirenz solution
- Sequence 2,3,1 (Experimental): Period A/ Visit 2: Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, homogenized to drug rich particles, oral administration (product 2) Period B/ Visit 6: Efavirenz solution, 3 mg, oral administration (product 3) Period C/ Visit 10: Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, oral administration (product 1)
  Interventions: Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz; Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz homogenized to drug rich particles; Drug: Efavirenz solution
- Sequence 3,1,2 (Experimental): Period A/ Visit 2: Efavirenz solution, 3 mg, oral administration (product 3) Period B/ Visit 6: Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, oral administration (product 1) Period C/ Visit 10: Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, homogenized to drug rich particles, oral administration (product 2)
  Interventions: Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz; Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz homogenized to drug rich particles; Drug: Efavirenz solution

INTERVENTIONS:
Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz — Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, oral administration (product 1)
Drug: Hot-melt extruded amorphous solid dispersion of Efavirenz homogenized to drug rich particles — Hot-melt extruded amorphous solid dispersion of Efavirenz, 50 mg, homogenized to drug rich particles, oral administration (product 2)
Drug: Efavirenz solution — Efavirenz solution, 3 mg, oral administration (product 3)

SUMMARY:
It is the aim of the study to investigate the functioning of a drug delivery system (drug-rich particles forming hot-melt extruded amorphous solid dispersions) with respect to mechanisms of bioavailability of poorly soluble drug substances.

DETAILED DESCRIPTION:
Poor drug solubility, and therefore low bioavailability, remains a problem in drug development that causes many drug candidates to drop out during drug development. Bioavailability is linked to drug solubility and intestinal permeability. A promising method to increase drug solubility, and therefore bioavailability, is the formulation of the drug as hot-melt extruded amorphous solid dispersion drug delivery systems, which have been shown to potentially increase in vivo and clinical bioavailability.The mechanisms that lead to increased bioavailability are not understood completely.

In this study, investigators investigate the role of amorphous solid dispersions and thereof generated drug-rich particles on bioavailability and their in vivo behaviour. Investigators do so by administering the delivery system at different stages in the process of drug availability.

Primary objectives are the pharmacokinetic analysis of a model formulation using efavirenz as model drug tracer in human.

* Comparison of pharmacokinetic parameters such as relative bioavailability and further parameters derived from pharmacokinetic analysis and corresponding interpatient variabilities.
* Mechanistic analysis of pharmacokinetic data, such as determination of in vivo dissolution from the solid formulation (study product 1) to drug rich particles (study product 2) using numerical deconvolution or analysis of the effect of drug rich particles on the absorption rate of Efavirenz in comparison to the solution of Efavirenz (study product 3).

Secondary objectives are the comparison of obtained pharmacokinetic profiles to existing data of a conventional formulation with respect to:

* Comparison of pharmacokinetic parameters such as relative bioavailability and further parameters derived from pharmacokinetic analysis and corresponding interpatient variabilities.
* Extrapolation investigation from in vitro to in vivo data.

Safety objectives are the recording of any side effects or tolerability issues of the investigational drug delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Full mental and legal capacity, ability and willingness to understand and comply to study interventions and restrictions and to communicate with study personnel.
* Informed Consent, documented by signature (Informed Consent Form).
* Physically and mentally healthy male participants, age of 18 to 50 years.
* Body mass index (BMI) of 18.0 to 29.9 kg/m2, systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50- 90 mmHg and heart rate (HR) 45-90 bpm, measured on the leading arm, after 5 minutes in supine position, Hemoglobin ≥ 11 g/dl at screening.
* Normal physical examination, vital signs, laboratory workup (clinical chemistry and hematology), and electrocardiogram (ECG) (in opinion of the principal investigator).
* Normal renal and liver function based on blood tests (in opinion of the investigator).
* Medical history that is in line with the eligibility criteria. (in opinion of the investigator).
* No other conditions or circumstances that might compromise compliance with the study protocol or the quality of retrieved data (in opinion of the investigator).

Exclusion Criteria:

* Any acute or chronic illness or other clinically relevant findings at screening.
* Any physical or mental disorder or circumstance at present or in medical history that could interfere with the participant's safety during the clinical trial or with the study objectives.
* Any regular drug treatment within the last two weeks or planned for the time of the study (exceptions possible in opinion of the investigator).
* At presence of irregular drug treatment before the study, planned for the time of the study or irregular/regular substitution of endogenous substances, minerals, or trace elements, the investigator decides on exclusion on an individual basis valuing the safety of the participant and the quality of retrieved data (e.g. interactions with Efavirenz). For minor to moderate painful conditions, such as headaches or abdominal discomfort, paracetamol up to 1 g every 6 hours is acceptable.
* Any intake of a substance known to induce or inhibit drug metabolizing enzymes or transport system enzymes relevant for Efavirenz (CYP 2B6 and CYP 3A4) within a period of less than 10 times the respective elimination half-life.
* Vaccination (active or passive) ≤ one month before screening.
* Presence or history of allergies (except for mild forms of hay fever).
* History of hypersensitivity reactions to medication.
* History or presence of eating disorders.
* Presence of contraindications to treatment with Efavirenz, namely less than 40 kg body weight, co-medication with voriconazole, paritaprevir, ritonavir, dasabuvir, simeprevir, and hypericum perforatum.any co-medication (also plant products), or any liver disease.
* Presence of warnings concerning the treatment with Efavirenz, namely severe skin irritations in the medical history, psychiatric symptoms in the medical history, convulsions in the medical history, hepatitis B or C, presence of osteonecrosis in the medical history, or dyslipidemia at present or in medical history.
* History or presence of smoking, alcohol drinking (>20 g alcohol per day), or drug abuse.
* Blood donation or significant blood loss within 4 weeks prior to screening
* Known or suspected non-compliance
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
AUC | before dosing and at time points 15 minutes, 30 minutes, 45 minutes, 60 minutes, followed by sampling at 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, and 72 hours after dosing
  Area under the curve in plasma concentration - time profiles of efavirenz after administration of the different study products.
Relative bioavailability | before dosing and at time points 15 minutes, 30 minutes, 45 minutes, 60 minutes, followed by sampling at 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, and 72 hours after dosing
  Ratio between areas under the curve.
Cmax | before dosing and at time points 15 minutes, 30 minutes, 45 minutes, 60 minutes, followed by sampling at 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, and 72 hours after dosing
  Maximal concentration in the plasma concentration - time profiles of efavirenz after administration of the different study products.
Tmax | before dosing and at time points 15 minutes, 30 minutes, 45 minutes, 60 minutes, followed by sampling at 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, and 72 hours after dosing
  Time of maximal concentration in the plasma concentration - time profiles of efavirenz after administration of the different study products.
ka | before dosing and at time points 15 minutes, 30 minutes, 45 minutes, 60 minutes, followed by sampling at 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, and 72 hours after dosing
  Absorption rate constant from the concentration in the Plasma concentration - time profiles of efavirenz after administration of the different study products.
In vivo dissolution | before dosing and at time points 15 minutes, 30 minutes, 45 minutes, 60 minutes, followed by sampling at 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, and 72 hours after dosing
  Calculation of in vivo dissolution of based on the numerical deconvolution of plasma concentration - time profiles of efavirenz after administration of the different study products.

SECONDARY OUTCOMES:
Number of adverse drug reactions | During inclusion into study (36 to 54 days)
  Incidence and severity (CTCAE Version 5) of adverse reactions (adverse event suspected to be related to investigational drug deliver system, expected or not expected) during the whole study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Krähenbühl, Prof. Dr., Principal Investigator — University of Basel, Department Biomedicine
Locations (1):
- Pharmaceutical Technology, University of Basel, Pharmazentrum, Basel, Switzerland

REFERENCES:
- [Result] Schittny A, Waldner S, Duthaler U, Vorobyev A, Abramovich R, Krahenbuhl S, Puchkov M, Huwyler J. Particle Forming Amorphous Solid Dispersions: A Mechanistic Randomized Pharmacokinetic Study in Humans. Pharmaceutics. 2021 Mar 17;13(3):401. doi: 10.3390/pharmaceutics13030401. PMID 33803049